CLINICAL TRIAL: NCT05071482
Title: Flumatinib Versus Imatinib Combined With Multiagent Chemotherapy for Newly Diagnosed Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia: A Prospective, Open-label，Randomized，Multi-center Clinical Trial
Brief Title: Flumatinib Versus Imatinib Combined With Chemotherapy for de Novo Ph+ ALL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021024
Record Dates: First submitted 2021-09-09; First posted 2021-10-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-05

CONDITIONS: Acute Leukemia
Keywords: acute lymphoblastic leukemia; flumatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — flumatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flumatinib arm (Experimental): 600 mg QD oral administration, fasting (2 hours before administration and 1 hour after administration).
  Interventions: Drug: Flumatinib
- imatinib arm (Active Comparator): 600 mg QD oral administration, with a meal
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Flumatinib — Flumatinib 600 mg qd will be given orally along with combination chemotherapy starting day 8 of induction chemotherapy. Flumatinib will be given continuously (if it's tolerable) for 2 years since achievement of complete remission (CR) as part of consolidation chemotherapy and maintenance therapy. Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT),or patients in whom MCR was achieved within 3 months after treatment and continued until transplantation can receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation and maintenance chemotherapy.
  Arms: flumatinib arm
Drug: Imatinib — Imatinib 600 mg qd will be given orally along with combination chemotherapy starting day 8 of induction chemotherapy. Imatinib will be given continuously (if it's tolerable) for 2 years since achievement of complete remission (CR) as part of consolidation chemotherapy and maintenance therapy. Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT),or patients in whom MCR was achieved within 3 months after treatment and continued until transplantation can receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation and maintenance chemotherapy.
  Arms: imatinib arm

SUMMARY:
Compared with patients with philadelphia chromosome-negative Acute Lymphoblastic Leukemia (Ph- ALL), patients with Ph-positive (Ph+) ALL exhibit a comparatively poor prognosis. Fortunately, significant improvements have been found in response rates, disease-free survival (DFS), and overall survival (OS) for patients with Ph+ ALL with the introduction of tyrosine kinase inhibitor (TKI) therapy to treatment regimens. Based on improvements in efficacy and tolerability, next-generation TKIs have been widely used in first-line treatment for chronic myeloid leukemia (CML). Flumatinib, a TKI with more potent binding affinity for BCR-ABL1 tyrosine kinase than imatinib, demonstrated higher rates of responses, faster and deeper responses in FESTnd trial, which suggested that flumatinib might show improved clinical efficacy for treating Ph+ ALL compared with imatinib. The investigators therefore hypothesized that the addition of flumatinib to combinatorial chemotherapy regimen would demonstrate greater efficacy compared with the prior use of imatinib in treating Ph+ ALL. This study explored the safety and efficacy of flumatinib versus imatinib when combined with multi-agent chemotherapy in patients with newly diagnosed Ph+ ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years, male or female;
2. Newly diagnosed Philadelphia chromosome positive(either t(9;22) and/or BCR-ABL positive and/ or FISH positive) acute lymphoblastic leukemia; Patients will be diagnosed according to morphologic,immunologic, cytogenetic and molecular(MICM) criteria, including bone marrow morphology, immunophenotype, cytogenetic and molecular genetic (BCR/ABL gene, qualitative and quantitative analysis) examination.
3. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2;
4. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤5 x ULN if leukemic involvement of the liver is present; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; normal electrolytes: Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN;
5. Cardiac color Doppler ultrasound ejection fraction ≥ 45%;
6. Subject has provided written informed consent prior to any screening procedure;

Exclusion Criteria:

1. Lymphoid blast crisis of chronic myelocytic leukemia (CML);
2. Previous or ongoing systemic anti-ALL therapy (including but not restricted to TKI and/or radiotherapy, except for appropriate pre-treatment);
3. Patients with clinical manifestations of central or extramedullary invasion of leukemia at diagnosis;
4. Identification of T315I mutation;
5. Concurrent participation in another clinical study with an investigational medical product;
6. Any concurrent severe and/or uncontrolled medical condition, which could, in the opinion of the investigator, compromise participation in the study;
7. History of neurological or psychiatric disorders, including epilepsy or dementia;
8. Major surgery within 4 weeks or failure to recover from previous surgery;
9. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention;
10. Female patients who are pregnant or breast feeding or patients of childbearing potential and male patients whose sexual partner(s) are women of childbearing potential not willing to use a highly effective method of contraception;
11. Clinically significant, uncontrolled or active cardiovascular disease, specifically including, but not restricted to: any history of myocardial infarction, stroke, or revascularization; unstable angina or transient ischemic attack within 6 months prior to enrolment; congestive heart failure within 6 months prior to enrolment or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards; history of clinically significant (as determined by the treating physician) atrial arrhythmia; any history of ventricular arrhythmia; any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism;Uncontrolled hypertension;
12. Active known positive HIV serology;
13. Active serious infection not controlled by oral or intravenous antibiotics;
14. Patients with known allergies or contraindications to the study drug;
15. Patients with bleeding disorders unrelated to ALL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Relapse free survival | up to 24 months
  From the date of complete remission(CR) until the date of documented relapse or death due to any cause or the last follow-up day

SECONDARY OUTCOMES:
The rate of adverse events | through study completion, up to 24 months
  The incidence and severity of neutropenia, anemia, rash, hypophosphatemia, edema, limb pain, and other adverse events.
The composite CR rate | up to 2 month
  Both CR and molecular CR are obtained at the end of induction
The complete remission (CR) rate，CRi rate and overall remission rate（ORR） | up to 2 month
The minimal residual disease (MRD) negative rate by Flow Cytometry (FCM) | up to 24 months
The molecular CR rate | up to 6 months
The rate of primary induction failure(PIF) | up to 6 months
The duration of molecular CR | up to 24 months
The duration of CR | up to 24 months
Time to treatment failure | up to 24 months
The cumulative recurrence rate | up to 24 months
The CNS recurrence rate | up to 24 months
Event free survival(EFS) | up to 24 months
Overall survival(OS) | up to 24 months
The rate of interruption and discontinuation due to AE | up to 24 months

OTHER OUTCOMES:
ABL kinase region mutation status at molecular relapse (MREL) and hematologic relapse (HREL) | up to 24 months
The plasma and cerebrospinal fluid (CSF) level of flumatinib | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China